CLINICAL TRIAL: NCT00006340
Title: A PHASE I TRIAL OF BUTYRATE AND GANCICLOVIR IN EBV-ASSOCIATED MALIGNANCIES
Brief Title: Ganciclovir Plus Arginine Butyrate in Treating Patients With Cancer or Lymphoproliferative Disorders Associated With the Epstein Barr Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Purpose: Treatment
Other Study IDs: CDR0000064947; BUMC-3756; BUSM-FDR001532; NCI-V00-1609
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Leukemia; Lymphoma; Precancerous Condition; Small Intestine Cancer
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; small intestine lymphoma; childhood immunoblastic large cell lymphoma; grade I lymphomatoid granulomatosis; grade II lymphomatoid granulomatosis; adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; childhood grade III lymphomatoid granulomatosis; recurrent childhood grade III lymphomatoid granulomatosis; recurrent grade I lymphomatoid granulomatosis; recurrent grade II lymphomatoid granulomatosis; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; T-cell large granular lymphocyte leukemia; stage II grade 1 follicular lymphoma; stage II grade 2 follicular lymphoma; stage II grade 3 follicular lymphoma; stage II adult diffuse small cleaved cell lymphoma; stage II adult diffuse mixed cell lymphoma; stage II adult diffuse large cell lymphoma; stage II adult immunoblastic large cell lymphoma; stage II adult lymphoblastic lymphoma; stage II adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage II mantle cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage II small lymphocytic lymphoma; stage II marginal zone lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precancerous Conditions; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Leukemia, Large Granular Lymphocytic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — arginine butyrate; Ganciclovir

INTERVENTIONS:
Drug: arginine butyrate
Drug: ganciclovir

SUMMARY:
RATIONALE: The Epstein Barr virus can cause cancer and lymphoproliferative disorders. Ganciclovir is an antiviral drug that acts against the Epstein Barr virus. Arginine butyrate may make virus cells more sensitive to ganciclovir. Combining ganciclovir and arginine butyrate may kill more Epstein Barr virus cells and tumor cells.

PURPOSE: Phase I trial to study the effectiveness of arginine butyrate plus ganciclovir in treating patients who have cancer or lymphoproliferative disorders that are associated with the Epstein Barr virus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety, toxicity, and the reversibility of toxicity of arginine butyrate in patients with Epstein Barr virus-induced malignancies or lymphoproliferative disorders.
* Determine the clinical pharmacology of arginine butyrate when administered with ganciclovir, including plasma half life and major routes of elimination in these patients.
* Determine the biologic effects of arginine butyrate in terms of inducing sensitivity to ganciclovir in tissue samples from selected patients.
* Determine the antitumor activity of this treatment regimen in these patients.

OUTLINE: Patients receive ganciclovir IV over 1 hour twice a day on days -1 to 21 for the first course (days 0-21 for all subsequent courses) and escalating doses of arginine butyrate IV continuously on days 0-21. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for a minimum of 42 days.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy or lymphoproliferative disease including the following:

  * Nasopharyngeal carcinoma
  * Hodgkin's lymphoma
  * African Burkitt's lymphoma
  * T-cell non-Hodgkin's lymphoma
  * B-cell non-Hodgkin's lymphoma if Epstein Barr Virus (EBV) positive
  * Other lymphomas associated with immunodeficiency or immunosuppression, including AIDS-related lymphoma
  * B-cell lymphoproliferative disorders
* Monoclonal or oligoclonal B-cell lymphoid disease (no polyclonal disease)
* EBV positive by immunohistochemistry or in situ hybridization

  * Negative serology for EBV allowed

PATIENT CHARACTERISTICS:

Age:

* 3 and over

Performance status:

* Any status

Hematopoietic:

* Absolute granulocyte count at least 1,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Aminotransferase less than 2 times normal

Renal:

* Creatinine less than 3.0 mg/dL
* Creatinine clearance greater than 30 mL/min

Cardiovascular:

* No acute myocardial infarction within the past 6 months
* No atrial fibrillation within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior bone marrow or stem cell transplantation allowed
* No concurrent immunotherapy
* No concurrent interferon or tacrolimus

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered
* No concurrent cytotoxic chemotherapy

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* Recovered from prior radiotherapy

Surgery:

* Not specified

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-12; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas V. Faller, MD, PhD, Study Chair — Boston Medical Center
Locations (6):
- United States (3):
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Hopital Necker, Paris, France
- Medizinische Hochschule Hannover, Hanover, Germany
- Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan, Italy

REFERENCES:
- [Background] Faller DV, Mentzer SJ, Perrine SP. Induction of the Epstein-Barr virus thymidine kinase gene with concomitant nucleoside antivirals as a therapeutic strategy for Epstein-Barr virus-associated malignancies. Curr Opin Oncol. 2001 Sep;13(5):360-7. doi: 10.1097/00001622-200109000-00008. PMID 11555713
- [Background] Mentzer SJ, Perrine SP, Faller DV. Epstein--Barr virus post-transplant lymphoproliferative disease and virus-specific therapy: pharmacological re-activation of viral target genes with arginine butyrate. Transpl Infect Dis. 2001 Sep;3(3):177-85. doi: 10.1034/j.1399-3062.2001.003003177.x. PMID 11493400
- [Result] Perrine SP, Hermine O, Small T, Suarez F, O'Reilly R, Boulad F, Fingeroth J, Askin M, Levy A, Mentzer SJ, Di Nicola M, Gianni AM, Klein C, Horwitz S, Faller DV. A phase 1/2 trial of arginine butyrate and ganciclovir in patients with Epstein-Barr virus-associated lymphoid malignancies. Blood. 2007 Mar 15;109(6):2571-8. doi: 10.1182/blood-2006-01-024703. Epub 2006 Nov 21. PMID 17119113
- [Result] Mentzer SJ, Fingeroth J, Reilly JJ, Perrine SP, Faller DV. Arginine butyrate-induced susceptibility to ganciclovir in an Epstein-Barr-virus-associated lymphoma. Blood Cells Mol Dis. 1998 Jun;24(2):114-23. doi: 10.1006/bcmd.1998.0178. PMID 9628848